CLINICAL TRIAL: NCT03278184
Title: The Role of Transcranial Direct Current Stimulation in Reduction of Pain and Postoperative Opioids Consumption After Spine Surgery, Double Blinded Study
Brief Title: Transcranial Direct Current Stimulation in Reduction of Pain and Postoperative Opioids Consumption After Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Saeid Metwaly Abouelyazid Elsawy, Assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: post tDCS
Record Dates: First submitted 2017-09-05; First posted 2017-09-11 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tDCS sham motor cortex (Sham Comparator): 25 participants will have sham stimulation for 20 minutes using transcranial direct current stimulation device.
  Interventions: Device: tDCS sham motor cortex
- Active motor cortex stimulation (Active Comparator): 25 participants will have active stimulation targeting the left motor cortex for 20 minutes using transcranial direct current stimulation device.
  Interventions: Device: active motor cortex stimulation
- active prefrontal cortex stimulation (Active Comparator): 25 participants will have active stimulation targeting the left dorsolateral prefrontal cortex for 20 minutes using transcranial direct current stimulation device.
  Interventions: Device: active prefrontal cortex stimulation

INTERVENTIONS:
Device: tDCS sham motor cortex — the intervention 25 participants will be subjected to spine surgery then participants will be subjected to sham stimulation targeting left motor cortex area using the transcranial direct current stimulation device for 30 seconds then stop for 20 minutes.
  Arms: tDCS sham motor cortex
Device: active prefrontal cortex stimulation — the intervention 25 participants will be subjected to spine surgery then participants will be subjected to an active stimulation targeting left dorsolateral prefrontal cortex area using the transcranial direct current stimulation device with a current intensity of 2 mA for 20 min
  Arms: active prefrontal cortex stimulation
Device: active motor cortex stimulation — the intervention 25 participants will be subjected to spine surgery then participants will be subjected to an active stimulation targeting left motor cortex area using the transcranial direct current stimulation device with a current intensity of 2 mA for 20 min
  Arms: Active motor cortex stimulation

SUMMARY:
The experience of pain derives from changes in brain excitability. Therefore, modulating the excitability of cortical areas involved in pain processing may become an attractive option in the context of multimodal analgesia during the postoperative period.

DETAILED DESCRIPTION:
The combination of analgesic drugs acting on different mechanisms can potentiate the effects of analgesia. Moreover, the understanding of pain physiology at the molecular level supports the development of new specific drugs. Indeed, new neurophysiological models of pain processing by the brain are becoming exquisitely refined and are supported by electrophysiological and functional brain imaging studies. One of the interesting concepts that stemmed from these studies is the evidence that the experience of pain is reflected in the central nervous system by widespread activations and excitability changes within a network of interconnected cortical areas and subcortical structures. The network processing of noxious information and their limbic and emotional consequences has been termed the "pain matrix." The continuous observation of the activity and excitability changes that parallel the pain experience led to the development of a new therapeutic approach: the use of central nervous system stimulation techniques.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent to participate in the study.
* postoperative spine surgery patients(discectomy and/or laminectomy).
* American society of anesthesiology scores I to II patients.

Exclusion Criteria: the participant who has any history of:

* an adverse reaction to brain stimulation.
* a seizure
* an unexplained loss of consciousness
* a stroke
* serious head injury
* surgery to their head
* any brain related, neurological illnesses
* any illness that may have caused brain injury
* frequent or severe headaches
* metal in your head (outside the mouth) such as shrapnel, surgical clips, or fragments from welding
* any implanted medical devices such as cardiac pacemaker's or medical pumps
* taking any analgesic medications in the past 24 hours
* pregnancy
* anyone in your family has epilepsy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
the total consumption of morphine administered by patients during the first two days postoperative | 48 hours postoperative
  the investigator will calculate the amount of morphine used during the first two days postoperative.

SECONDARY OUTCOMES:
Pain severity assessment using visual analogue scale (VAS score from 0-10) | 30 minutes after every sessions and at the third day
  the investigator will assess the pain at base line and at the end of sessions
HADS score | before surgery and at the third day
  hospital anexiety and depression score

CONTACTS AND LOCATIONS:
Overall Officials: Saeid M Elsawy, MBBch, Principal Investigator — Assiut University
Locations (2):
- Saeid Metwaly Elsawy, Asyut, Egypt
- Saeid Elsawy, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided